CLINICAL TRIAL: NCT06013241
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of the Efficacy and Safety of Brensocatib in Participants With Chronic Rhinosinusitis Without Nasal Polyps - The BiRCh Study
Brief Title: A Study of the Efficacy and Safety of Brensocatib in Participants With Chronic Rhinosinusitis Without Nasal Polyps (CRSsNP)
Acronym: BiRCh
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INS1007-221; 2022-502481-24-00 (Other: EU CT Number)
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Chronic Rhinosinusitis Without Nasal Polyps
Keywords: CRSsNP
MeSH Terms: interventions — brensocatib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Brensocatib 40 mg (Experimental): Participants will receive brensocatib 40 mg tablet, orally, QD for 24 weeks along with mometasone furoate nasal spray (MFNS) by nasal route as background therapy at a stable dose according to the Investigator's discretion and local guidance.
  Interventions: Drug: Brensocatib; Drug: Mometasone furoate nasal spray (MFNS)
- Brensocatib 10 mg (Experimental): Participants will receive brensocatib 10 mg tablet, orally, QD for 24 weeks along with MFNS by nasal route as background therapy at a stable dose according to the Investigator's discretion and local guidance.
  Interventions: Drug: Brensocatib; Drug: Mometasone furoate nasal spray (MFNS)
- Placebo (Placebo Comparator): Participants will receive a brensocatib-matching placebo tablet, orally, QD for 24 weeks along with MFNS by nasal route as background therapy at a stable dose according to the Investigator's discretion and local guidance.
  Interventions: Drug: Placebo; Drug: Mometasone furoate nasal spray (MFNS)

INTERVENTIONS:
Drug: Brensocatib — Film-coated tablet.
  Other Names: INS1007
  Arms: Brensocatib 10 mg; Brensocatib 40 mg
Drug: Placebo — Film-coated tablet.
  Arms: Placebo
Drug: Mometasone furoate nasal spray (MFNS) — Nasal spray suspension.

SUMMARY:
The primary purpose of the study is to evaluate the efficacy of brensocatib at 10 and 40 milligrams (mg) once daily (QD) compared with placebo in improving clinical symptoms of CRSsNP.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have at least a 12-week history before Screening Visit of CRSsNP and confirmed by endoscopy at Visit 1 (Screening).
* Participants must have a NCS of ≥2 at Visit 1 (Screening Visit) and Visit 2 (Baseline; average score in the week prior to randomization).
* Participants must have sTSS (nasal congestion [NC], anterior/posterior rhinorrhea, facial pain/pressure) ≥5 at Visit 1 (Screening) and at Visit 2 (Baseline; average score in the week prior to randomization).
* Participants who have at least 1 of the 3 following features:

  1. Previous sinonasal surgery for CRS, including but not limited to fenestrated endoscopic sinus surgery and balloon sinuplasty.
  2. Received medical treatment with systemic corticosteroids (SCS) to treat symptoms of CRS as defined by any dose and duration within 1 year of Screening Visit or intolerance/contraindication to SCS.
  3. Received a course of antibiotics to treat symptoms of CRS within 1 year before the Screening Visit.
* Participants who have a blood eosinophil count ≤750 cells/microliter (μL) at Visit 1 (Screening).
* Participants who have bilateral inflammation of paranasal sinuses in the CT scan performed during Screening and bilateral ethmoid and/or maxillary opacification before randomization as confirmed by the central reader.
* Participants who have a SNOT-22 score of ≥20 at Visit 1 (Screening) and Visit 2 (Baseline).
* Participants who have received a stable daily dose regimen of MFNS for at least 4 weeks before Visit 2 (Baseline).

Exclusion Criteria:

* Diagnosis of unilateral or bilateral chronic rhinosinusitis with nasal polyps (CRSwNP).
* Clinical diagnosis of cystic fibrosis (CF) or primary ciliary dyskinesia.
* Scheduled sinus surgery at any time during the study.
* Participants who have had nasal surgery within 4 weeks before Visit 1 (Screening) and during the Screening Period.
* Significant oral maxillofacial structural abnormalities or severe septal deviation.
* Participants with radiological suspicion or confirmed invasive fungal rhinosinusitis, odontogenic sinusitis, osteomas, or nasal tumors.
* Participants with acute change in symptoms consistent with acute rhinosinusitis.
* Participants with seasonal allergic rhinitis whose symptoms coincide with the treatment period of the study.
* Participants with moderate to severe atopic dermatitis requiring treatment with high potency topical steroids or topical calcineurin inhibitors or biologics.
* Clinical diagnosis of Papillon-Lefèvre syndrome.

Note: Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Change From Baseline to the 28-day Average of Daily Sinus Total Symptom Score (sTSS) at Week 24 | Baseline and Week 24

SECONDARY OUTCOMES:
Change From Baseline in Percentage of Sinus (Maxillary and Ethmoid) Opacification as Measured by Volumetry at Week 24 | Baseline and Week 24
  The computed tomography (CT) scan performed during Screening (considered as Baseline) and at Week 24 will be used for the volumetric assessment of maxillary and ethmoid sinus opacification.
Change From Baseline in Modified Lund-MacKay (LMK) Computed Tomography (CT) Score at Week 24 | Baseline and Week 24
Proportion of Participants Requiring Rescue (Antibiotics, Systemic Corticosteroids [SCS], and/or Nasal Surgery) due to Worsening of any Chronic Rhinosinusitis (CRS) Symptoms up to Week 24 | Baseline up to Week 24
Change From Baseline to the 28-day Average of Daily Nasal Congestion Score (NCS) at Week 24 | Baseline and Week 24
Change From Baseline to the 28-day Average of Daily Peak Nasal Inspiratory Flow (PNIF) at Week 24 | Baseline and Week 24
Change From Baseline in Sino-Nasal Outcome Test (SNOT-22) Total Score at Week 24 | Baseline and Week 24
Plasma Concentration of Brensocatib | Pre-dose and at multiple timepoints post-dose up to Week 24
Percentage of Participants who Experienced at Least One Adverse Event (AE) | Up to 28 weeks
  Determination of the safety and tolerability of brensocatib compared with placebo.

CONTACTS AND LOCATIONS:
Locations (100):
- United States (27):
  - USA034, Tucson, Arizona
  - USA002, Roseville, California
  - USA006, Upland, California
  - USA016, Boca Raton, Florida
  - USA019, Hollywood, Florida
  - USA001, Miami, Florida
  - USA009, Tampa, Florida
  - USA031, Chicago, Illinois
  - USA021, Chicago, Illinois
  - USA003, New Albany, Indiana
  - USA035, Mandeville, Louisiana
  - USA026, Baltimore, Maryland
  - USA011, Columbia, Missouri
  - USA024, St Louis, Missouri
  - USA033, New York, New York
  - USA028, Tulsa, Oklahoma
  - USA004, Tulsa, Oklahoma
  - USA015, Hershey, Pennsylvania
  - USA023, Charleston, South Carolina
  - USA022, North Charleston, South Carolina
  - USA025, Dallas, Texas
  - USA037, Fredericksburg, Texas
  - USA029, Houston, Texas
  - USA018, Houston, Texas
  - USA030, San Antonio, Texas
  - USA038, Tomball, Texas
  - USA005, Norfolk, Virginia
- Argentina (17):
  - ARG015, La Plata, Buenos Aires
  - ARG001, La Plata, Buenos Aires
  - ARG006, Lobos, Buenos Aires
  - ARG005, Buenos Aires, Ciudad Autónoma de BuenosAires
  - ARG012, Buenos Aires, Ciudad Autónoma de BuenosAires
  - ARG011, Buenos Aires, Ciudad Autónoma de BuenosAires
  - ARG017, Buenos Aires, Ciudad Autónoma de BuenosAires
  - ARG013, San Rafael, Mendoza Province
  - ARG007, Rosario, Santa Fe Province
  - ARG010, Rosario, Santa Fe Province
  - ARG004, Rosario, Santa Fe Province
  - ARG009, San Miguel de Tucumán, Tucumán Province
  - ARG002, Mar del Plata
  - ARG014, Mendoza
  - ARG003, Mendoza
  - ARG016, Rosario
  - ARG008, Santa Fe
- Australia (2):
  - AUS001, Herston, Queensland
  - AUS002, Spearwood, Western Australia
- Belgium (3):
  - BEL001, Ghent, Oost-Vlaanderen
  - BEL002, Erpent
  - BEL003, Woluwe-Saint-Lambert
- Bulgaria (3):
  - BGR005, Sofia, Sofia-Grad
  - BGR003, Plovdiv
  - BGR006, Stara Zagora
- Canada (6):
  - CAN003, Vancouver, British Columbia
  - CAN006, London, Ontario
  - CAN007, Toronto, Ontario
  - CAN005, Montreal, Quebec
  - CAN001, Québec, Quebec
  - CAN002, Québec
- Czechia (4):
  - CZE002, Olomouc, Olomoucký kraj
  - CZE003, Pardubice, Pardubický kraj
  - CZE005, Nový Hradec Králové
  - CZE004, Prague
- Denmark (4):
  - DNK004, Hillerød, Capital
  - DNK001, København Ø, Capital
  - DNK003, Aarhus C, Central Jutland
  - DNK002, Køge, Zeeland
- France (4):
  - FRA002, Strasbourg, Bas-Rhin
  - FRA003, Marseille, Bouches-du-Rhône
  - FRA001, Nantes, Loire-Atlantique
  - FRA004, La Roche-sur-Yon, Vendée
- Germany (7):
  - GER004, Wiesbaden, Hesse
  - GER009, Leipzig, Saxony
  - GER003, Mittweida, Saxony
  - GER008, Lübeck, Schleswig-Holstein
  - GER005, Jena, Thuringia
  - GER007, Berlin
  - GER001, Dresden
- HUN003, Pécs, Baranya, Hungary
- Italy (3):
  - ITA001, Rozzano, Lombardy
  - ITA002, Sassari, Sardinia
  - ITA003, Pisa, Tuscany
- Poland (10):
  - POL002, Poznan, Greater Poland Voivodeship
  - POL010, Poznan, Greater Poland Voivodeship
  - POL005, Krakow, Lesser Poland Voivodeship
  - POL007, Wieliczka, Lesser Poland Voivodeship
  - POL009, Wroclaw, Lower Silesian Voivodeship
  - POL003, Lublin, Lublin Voivodeship
  - POL001, Warsaw, Masovian Voivodeship
  - POL004, Bialystok, Podlaskie Voivodeship
  - POL006, Katowice, Silesian Voivodeship
  - POL008, Warsaw
- Portugal (5):
  - PRT001, Guimarães, Braga District
  - PRT003, Lisbon, Lisbon District
  - PRT005, Senhora da Hora, Porto District
  - PRT004, Aveiro
  - PRT002, Braga
- Spain (4):
  - ESP003, Santander, Cantabria
  - ESP002, Jerez de la Frontera, Cádiz
  - ESP004, Málaga, Málaga
  - ESP001, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Prescreening tool — https://connect.trialscope.com/studies/745d2e53-fe55-4723-a23a-e932a8858951